## NCT02914119

Use of Neuromuscular Blocking Agents and Neuromuscular Monitoring in 7 Danish Teaching Hospitals 03 August 2019

## Statistical analyses

Continuous variables and ordinal variables are presented as mean (SD) or median (inter-quartile range (IQR)), categorical variables as number (percentage). Analyses were performed using SPSS version 22 and 25 (IBM Corporation, USA).